CLINICAL TRIAL: NCT05904899
Title: An Evaluation of the Implementation of the Care and Monitoring at Home Program- A New Paradigm for Acute Care Management of Cancer Patients
Status: Suspended | Type: Observational
Why Stopped: PI Request
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-1034; NCI-2023-04326 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To understand the experience of patients receiving care in the Care and Monitoring at Home program at MD Anderson. Researchers intend to use this information to study and possibly improve the hospital care at home program.

DETAILED DESCRIPTION:
OBJECTIVES

Primary Objectives

The objective of this observational study is to assess the feasibility of providing hospital substitution hospital level care in the home for patients with cancer through the CaMH Program. Our primary gauge of feasibility will be a care escalation rate of <20%, defined as the proportion of patients who initiate care in our HaH program but are transferred back to the inpatient setting to complete the care episode. This threshold is consistent with the published literature.15 In addition, a "feasible" designation will require a median score > 3 on each of three post-discharge survey implementation measures - the Feasibility of Implementation Measure, Acceptability of Implementation Measure, and Intervention Appropriateness Measure.

Secondary Objectives

Secondary objectives will include patient experience and perception about CaMH, length of stay, rate of clinical adverse events during CaMH (falls, pressure ulcers, medication errors) and 30-days after discharge, 7-day readmission, 30-day readmission, and 30-day emergency department visit rate. (Note, the aforementioned adverse events could occur as a result of participation in CaMH. However, minimal adverse events are expected a result of participation in this observational study (see adverse events below)). A patient will be considered to have an ER visit or hospital readmission if these events are documented in the medical record OR the patient reports the event on the survey.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be eligible for enrollment in this study if they have accepted enrollment in CaMH. No patients will be excluded if they are enrolled in CaMH.
* Cognitively impaired adults will be able to participate in the study if an adults proxy provides informed consent and completes survey materials on their behalf.

Exclusion Criteria:

- Children and pregnant women will not be enrolled in the CaMH program, and therefore not eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants enrolled in the Care and Monitoring at Home program at MD Anderson.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life questionnaires (QOL) | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Josiah Halm, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org